CLINICAL TRIAL: NCT02607410
Title: Short and Long Term Effects of a Dypeptidil-peptidase-4 Versus Bedtime NPH Insulin as add-on Therapy in Patients With Type 2 Diabetes
Brief Title: Sitagliptin (DPP-4 Inhibitor) and NPH Insulin in Patients With T2D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Maria Elizabeth Rossi da Silva, MD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERS2015
Record Dates: First submitted 2015-11-06; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; sitagliptin; NPH insulin; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors; Insulin, Isophane; Insulin, Long-Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sitagliptin (Active Comparator): 100mg every day of sitagliptin in patients that were previosly using metformin and glyburide
  Interventions: Drug: sitagliptin
- NPH insulin (Active Comparator): NPH insulin will be applied bedtime every night in patients that awere previously using metformin and glyburide,The insulin dosage will be adjusted to fasting glycemia between 90 and 100 mg / dL
  Interventions: Drug: NPH insulin

INTERVENTIONS:
Drug: sitagliptin — patients with type 2 diabetes,inadequately controlled with metformin plus glyburide, HbA1c between 6.6 to 10%, will be randomized to the addition of sitagliptin (Sitagliptin Group) or of bedtime NPH insulin (NPH Group) during one year
  Other Names: DPP-4 inhibitor
  Arms: sitagliptin
Drug: NPH insulin — patients with type 2 diabetes,inadequately controlled with metformin plus glyburide, HbA1c between 6.6 to 10%, will be randomized to the addition of sitagliptin (Sitagliptin Group) or of bedtime NPH insulin (NPH Group) during one year
  Other Names: long-acting insulin
  Arms: NPH insulin

SUMMARY:
To compare the short and long term effects of inhibitor of the DPP-IV enzyme, sitagliptin , with bedtime NPH insulin in patients with T2D inadequately controlled with sulphonylurea plus biguanide: effects on beta cell function and on metabolic profile.

DETAILED DESCRIPTION:
Glucose control is fundamental in the treatment of type 2 diabetes (DM2). Studies suggest that drugs that boost levels of glucagon-like peptide (GLP-1) improve glycemic control and have long-term beneficial effect on the function of pancreatic beta cells. Objective: To compare the short and long term effects of sitagliptin (which inhibits the DPP-IV enzyme, increasing the levels of GLP-1) with bedtime NPH insulin in patients with T2D inadequately controlled with sulphonylurea plus biguanide. Effects on beta cell function and on metabolic profile were analyzed. Methods: 40 patients with DM2, HbA1c between 6.6 to 10%, in use of metformin and glibenclamide will be randomized to the addition of sitagliptin (Sitagliptin Group) or of bedtime NPH insulin (NPH Group). Measurements of HbA1c, metabolic and hormonal profile at fasting and post-meal (every 30 minutes for 4 hours) will be evaluated before and after 6 months (short term) and 12 months (long term) of adding sitagliptin or NPH insulin.

ELIGIBILITY:
Inclusion Criteria

* outpatients with T2D inadequately controlled with metformin plus glyburide
* HbA1c levels between 6.6 and 10%
* body mass index < 35 kg/m2

Exclusion Criteria

* heart failure
* respiratory failure
* uncontrolled hypertension
* impaired hepatic function
* impaired reanl function
* endocrine disorder
* gastrointestinal disorder
* malignancy
* alcohol abuse
* previous use of insulin
* previou use of based incretin therapy
* type 1 diabetes.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
improvement in HbA1c levels | six and twelve months
  Changes in fasting blood levels of HBA1c (%)

SECONDARY OUTCOMES:
improvement of beta cell function with a meal test | six and twelve months after each therapy at times zero, 30, 60, 120 and 180 minutes after meal test
  Changes in serum C-peptide levels (ng/mL)
improvement on alpha cell function with a meal test | six and twelve months after each therapy at times zero, 30, 60, 120 and 180 minutes after meal test
  Changes in plasma glucagon levels (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Maria ER Siva, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Muscelli E, Casolaro A, Gastaldelli A, Mari A, Seghieri G, Astiarraga B, Chen Y, Alba M, Holst J, Ferrannini E. Mechanisms for the antihyperglycemic effect of sitagliptin in patients with type 2 diabetes. J Clin Endocrinol Metab. 2012 Aug;97(8):2818-26. doi: 10.1210/jc.2012-1205. Epub 2012 Jun 8. PMID 22685234
- [Background] Aulinger BA, Bedorf A, Kutscherauer G, de Heer J, Holst JJ, Goke B, Schirra J. Defining the role of GLP-1 in the enteroinsulinar axis in type 2 diabetes using DPP-4 inhibition and GLP-1 receptor blockade. Diabetes. 2014 Mar;63(3):1079-92. doi: 10.2337/db13-1455. Epub 2013 Dec 2. PMID 24296715
- [Background] Retnakaran R, Qi Y, Opsteen C, Vivero E, Zinman B. Initial short-term intensive insulin therapy as a strategy for evaluating the preservation of beta-cell function with oral antidiabetic medications: a pilot study with sitagliptin. Diabetes Obes Metab. 2010 Oct;12(10):909-15. doi: 10.1111/j.1463-1326.2010.01254.x. PMID 20920044